CLINICAL TRIAL: NCT06799819
Title: Impact of Free Mobility on FDG Uptake During a PET Scan: Randomized Controlled Non-inferiority Study
Brief Title: Impact of Free Mobility on FDG Uptake in PET Scans
Acronym: MOBITEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHUO-2024-16
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms; Whole Body Imaging
Keywords: FDG PET; muscular uptake; image quality; Diagnostic Technics and Procedures
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, comparative, single-center, non-inferiority and single-blind (for the evaluator) study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blind analysis of the imaging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobility group (Experimental): Participant will benefit from the study procedure (free mobility after FDG injection)
  Interventions: Behavioral: Mobility group
- Control group (No Intervention): participant will benefit from the standard examination procedure (rest after FDG injection)

INTERVENTIONS:
Behavioral: Mobility group — Free mobility between FDG injection and scanning (without exiting the Nuclear Medicine Department)
  Arms: Mobility group

SUMMARY:
Positron Emission Tomography (PET) is a rather long examination (around 2 hours), involving an injection of 18F-Fluorodeoxyglucose (FDG), which requires the patient to rest for 1 hour between the injection and the start of imaging. Some hospitals allow the patient to sit, read or use the telephone, but none allow the patient to move freely after injection, hence the interest of this work. The aim of this study is to demonstrate that free mobilization of the patient following 18F-FDG injection does not result in any significant difference in imaging quality (particularly muscular fixations), and therefore a medical interpretation identical to that of a patient who remains at rest.

DETAILED DESCRIPTION:
FDG-PET is a fairly long scan involving an injection of 18F-FDG. Because of the fear of muscular fixations, the guidelines recommend for rest between injection and image acquisition. Indeed, some studies have demonstrated significant muscular uptake of the radiopharmaceutical in the event of major muscular effort prior to the examination. However, to investigators knowledge, the effect of free mobilization between injection and scan has not been evaluated. The aim of this study is to demonstrate that free mobilization of the participant after 18F-FDG injection does not result in a significant difference in imaging quality (especially muscular fixation) and therefore in a medical interpretation identical to that of a patient who remains at rest. Investigators also want to assess the impact on participant comfort and stress.

Each participant will receive an information leaflet with his or her examination appointment. On arrival in the department, after the study has been explained by the investigator and the participant has had all his questions answered, participant may accept inclusion by signing a consent form or refuse it. Once the inclusion of the participant has been validated, the randomisation will be done: the control group will benefit from the standard examination procedure (rest after FDG injection) and the experimental group will benefit from the study procedure (free mobility after FDG injection). The participant will complete a questionnaire on level of stress and comfort after the imaging procedure, and the nuclear physician will provide a blind interpretation.

A review of all blinded examinations will be carried out by two nuclear physicians to establish an examination quality score.

An intermediate analysis will be carried out when 50% of exclusions have been reached to stop the study if the management studied is detrimental compared with standard management.

ELIGIBILITY:
Inclusion Criteria:

1. Adults
2. Patient referred for FDG PET (excluding brain PET) and carried out on an outpatient basis.

Exclusion Criteria:

1. Bedridden patients
2. Protected person (under guardianship or curatorship)
3. Persons under court protection
4. Persons deprived of liberty
5. Persons not affiliated to a social security scheme
6. Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Visual image quality score (in terms of muscle fixations) | Day 0
  The visual quality of the images will be the main evaluation criterion.
  An overall examination quality score will be given by the investigator for each patient, using a 3-point Likert scale:
  1. no muscular fixation (interpretable examination)
  2. some muscular fixations that do not interfere with medical interpretation (interpretable examination)
  3. significant muscular fixations that make the examination uninterpretable. The main evaluation criterion will be the proportion of score 1 in the two groups of patients (with and without strict rest), bearing in mind that images scored 3 are very rare.

SECONDARY OUTCOMES:
Cervical SUV max | Day 0
Lumbosacral SUV max | Day 0
Improving patient comfort | Day 0
  Item-by-item comparisons are made between the two groups
Level of stress | Day 0
  Item-by-item comparisons are made between the two groups
Examination quality score | Day 0
  Factors that may influence the examination quality score will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline FRAT, Principal Investigator — CHU Orléans
Locations (1):
- Centre Hospitalier Universitaire d'Orléans, Orléans, France

REFERENCES:
- [Background] Reinking MF, Osman MM. Prospective evaluation of physiologic uptake detected with true whole-body 18F-FDG PET/CT in healthy subjects. J Nucl Med Technol. 2009 Mar;37(1):31-7. doi: 10.2967/jnmt.108.055004. Epub 2009 Feb 17. PMID 19223428
- [Background] Karunanithi S, Soundararajan R, Sharma P, Naswa N, Bal C, Kumar R. Spectrum of Physiologic and Pathologic Skeletal Muscle (18)F-FDG Uptake on PET/CT. AJR Am J Roentgenol. 2015 Aug;205(2):W141-9. doi: 10.2214/AJR.14.13457. Epub 2015 May 22. PMID 26001118
- [Background] Tashiro M, Fujimoto T, Itoh M, Kubota K, Fujiwara T, Miyake M, Watanuki S, Horikawa E, Sasaki H, Ido T. 18F-FDG PET imaging of muscle activity in runners. J Nucl Med. 1999 Jan;40(1):70-6. PMID 9935060
- [Background] Okuyama C, Kusano K, Ito M, Takase A, Goda S, Kagawa S. Characteristic Muscular FDG Uptake Patterns Related to the Transportation Means Used by Patients to Visit the Hospital. Clin Nucl Med. 2023 Jun 1;48(6):549-552. doi: 10.1097/RLU.0000000000004622. Epub 2023 Mar 16. PMID 36928161
- [Background] Wang Y, Shao F, Zhang L, Luo X, Chen Y. Increased 18F-FDG Uptake in Multiple Muscles in a Patient With Violent Cough. Clin Nucl Med. 2017 Jun;42(6):451-453. doi: 10.1097/RLU.0000000000001655. PMID 28368886
- [Background] Vock J, Juengling FD, Krause T, Wissmeyer M. Muscular FDG uptake after chewing chewing gum in a patient with Hodgkin disease. Clin Nucl Med. 2007 Feb;32(2):124-7. doi: 10.1097/01.rlu.0000252337.14196.ed. No abstract available. PMID 17242567